CLINICAL TRIAL: NCT02769741
Title: A Randomized, Controlled-Feeding, Crossover Study to Assess the Effect of Cashews on Fasting Lipoprotein Levels
Brief Title: A Controlled-Feeding Study to Assess the Effect of Cashews on Fasting Lipoprotein Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kraft Heinz Company (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: BIO-1509
Record Dates: First submitted 2016-05-06; First posted 2016-05-12 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Volunteers
Keywords: Cashew; Lipoprotein

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crossover 1: Control Diet followed by Active Diet (Other): Treatment Period 1: Controlled diet without cashew nuts; Treatment Period 2: Controlled diet with cashew nuts
  Interventions: Other: Control followed by Cashews
- Crossover 2: Active Diet followed by Control Diet (Other): Treatment Period 1: Controlled diet with cashew nuts; Treatment Period 2: Controlled diet without cashew nuts
  Interventions: Other: Cashews followed by Control

INTERVENTIONS:
Other: Cashews followed by Control — Participants will receive the active diet with cashew nuts as a daily snack during Test Period I at a calorie level to achieve weight maintenance, and with a macronutrient composition representative of a typical diet for 28 days. Following a 14-day washout period, subjects will receive the control diet at the same calorie level, but with a control snack instead of cashew nuts during Test Period II.
  Arms: Crossover 2: Active Diet followed by Control Diet
Other: Control followed by Cashews — Participants will receive a controlled diet without cashew nuts during Test Period I at a calorie level to achieve weight maintenance, and with a macronutrient composition representative of a typical diet for 28 days. Following a 14-day washout period, subjects will receive the active diet at the same calorie level, but with cashew nuts as a daily snack during Test Period II.
  Arms: Crossover 1: Control Diet followed by Active Diet

SUMMARY:
This study will assess the nutritional effect of cashews on LDL-C concentrations and secondarily on other aspects of the fasting lipoprotein lipid profile in healthy men and women with moderately elevated cholesterol.

DETAILED DESCRIPTION:
This trial will utilize a randomized, two-period crossover design to examine the effects of cashew consumption on LDL-C and other aspects of the fasting lipoprotein lipid profile in healthy, moderately hyper-cholesterolemic individuals consuming a typical "American diet." Two arms consisting of two 28-day controlled-feeding treatment periods will allow for an isocaloric comparison of a diet with or without cashews.

ELIGIBILITY:
Inclusion Criteria:

* BMI of ≥18.00 and ≤32.00 kg/m^2
* Fasting LDL-C level ≥130 mg/dL and <200 mg/dL
* Fasting TG ≤350 mg/dL

Exclusion Criteria:

* CHD or CHD risk equivalent
* Pregnancy
* Use of lipid altering medications which cannot be stopped
* Certain liver, kidney, lung, or gastrointestinal conditions
* Poorly controlled hypertension
* Certain medications
* Allergy or sensitivity to nuts or other food/beverage or food/beverage component
* Active cancers treated within prior 2 years (except non-melanoma skin cancer)
* Significant weight loss or gain within prior 3 months

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in LDL-C concentration measured in blood | % change from baseline (day 0) to the end of the test period (day 28) for Test Period I and II.

SECONDARY OUTCOMES:
Total cholesterol change | % change from baseline (day 0) to the end of the test period (day 28) for Test Period I and II.
HDL-cholesterol change | % change from baseline (day 0) to the end of the test period (day 28) for Test Period I and II.
Non-HDL-cholesterol change | % change from baseline (day 0) to the end of the test period (day 28) for Test Period I and II.
Triglyceride change | % change from baseline (day 0) to the end of the test period (day 28) for Test Period I and II.
Total cholesterol/HDL-cholesterol ratio change | % change from baseline (day 0) to the end of the test period (day 28) for Test Period I and II.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lawless, MD, Principal Investigator — BioFortis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mah E, Schulz JA, Kaden VN, Lawless AL, Rotor J, Mantilla LB, Liska DJ. Cashew consumption reduces total and LDL cholesterol: a randomized, crossover, controlled-feeding trial. Am J Clin Nutr. 2017 May;105(5):1070-1078. doi: 10.3945/ajcn.116.150037. Epub 2017 Mar 29. PMID 28356271